CLINICAL TRIAL: NCT06659315
Title: Addressing Perinatal Depression and PMTCT Adherence in Malawi: A Couple-Based Approach
Brief Title: Prevention of Mother-to-child Transmission (PMTCT) Among Women Experiencing Depression in Malawi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Invest in Knowledge Initiative (IKI) - Zomba, Malawi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-40685; R34MH134725 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: HIV Antiretroviral Therapy (ART) Adherence; Perinatal Mental Health; Depression During Pregnancy; PMTCT
Keywords: Perinatal depression; Couples; Problem-solving; PMTCT; ART adherence

STUDY DESIGN:
Intervention Model Description: Couples will be randomized 1:1 to intervention or control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (No Intervention): Standard of care, e.g., regular HIV care, regular perinatal care, referrals to services for depression
- Couple-based problem solving (Experimental): A couples-based intervention to support perinatal women who are experience symptoms of depression. We will adapt the WHO Problem Management Plus manual for this study. There are 5 sessions that deal with stress management, problem-solving, behavioral activation, and skills to strengthen social support. The final session will be modified to enhance couple communication skills. Because many of our participants will be dealing with food scarcity, we will develop a priori strategies to help couple brainstorm dealing with this issue.
  Interventions: Behavioral: Couples Problem Solving Therapy

INTERVENTIONS:
Behavioral: Couples Problem Solving Therapy — A couples-based problem solving program to deal with depression, PMTCT adherence, and couple communication.
  Arms: Couple-based problem solving

SUMMARY:
Prevention of mother-to-child transmission (PMTCT) of HIV virtually eliminates transmission of HIV from mothers to their infants. Adherence to PMTCT (i.e., to antiretroviral therapy, infant prophylaxis, and exclusive breastfeeding) during pregnancy and the postpartum period is challenging, with evidence from sub-Saharan Africa (SSA) showing suboptimal adherence and persistent viremia among perinatal women. Perinatal depression (PD) is a major driver of women's poor adherence to PMTCT. Interventions that involve male partners to provide social and food/economic support could be a promising approach for addressing PD and PMTCT, yet few interventions have intervened with couples to improve systems of support, communication, and other dyadic processes. The investigators propose to develop and test a couple-based approach to intervene on the mother's perinatal depressive symptoms and to strengthen the relationship and support system for partners to work together around depression to improve PMTCT adherence. The study will take place in antenatal and HIV care settings in Zomba, Malawi. The specific aims are: (1) to develop a couple-based intervention to target perinatal depression (PD) based on an evidence-based approach using problem-solving therapy (PST), augmented with content on couple communication and problem-solving skills; and (2) to assess the feasibility and acceptability (F&A) of the intervention via a pilot randomized controlled trial (RCT). Our short-term goal is the produce a couple-focused PST intervention that can be added to the global health toolkit for treating depression in perinatal women. Our long-term goal is to produce a high-impact and sustainable intervention leveraging the couple relationship that can be scaled-up to address depression, PMTCT adherence, and family health.

DETAILED DESCRIPTION:
Although prevention of mother-to-child transmission of HIV (PMTCT) services are widely available, 140,000 infants contracted HIV in 2021 and the majority were in sub-Saharan Africa (SSA). Urgent attention is needed to address poor engagement in PMTCT care with more than half of mothers disengaged from care by six months postpartum. Perinatal depression (PD) is a robust predictor of poor engagement in HIV care and suboptimal PMTCT adherence-defined as adherence to antiretroviral therapy (ART), infant prophylaxis and testing, and exclusive breastfeeding. Few PD interventions have been developed to address PMTCT in SSA and none have involved male partners, who are often major sources of financial and emotional support. Nor have interventions targeted the couple dynamics that can influence the mother's experience of PD and ability to access PMTCT. This project aims to fill this gap by developing and evaluating a problem-solving therapy (PST) intervention with perinatal women and their male partners to reduce PD symptoms and improve adherence to PMTCT in Malawi.

Pregnancy and postpartum are challenging times for couples with the stress of a new child, rising food expenses and nutritional demands, potential for couple conflict with new stressors, and less opportunity for connection and intimacy-all of which are amplified in the presence of PD. Among perinatal women with HIV in Kenya, investigators found that women's mental health and adherence to PMTCT was worsened by intimate partner violence (IPV) but positively affected by social support from partners, including food support during pregnancy and the breastfeeding period. In Malawi, investigators found that women in higher functioning relationships (e.g., better intimacy, communication) reported lower levels of depression, whereas women who reported IPV had higher rates of depression. Together, this suggests that dyadic processes such as support, conflict, and communication are central for women's experience of depression and for PMTCT. However, most PD interventions have focused on women alone rather than the dyad, which may explain why half of women treated for PD have reoccurring symptoms.

In this study, the investigators propose a couple-based intervention to strengthen couple relationships and support for partners to work together around depression, food insecurity, and PMTCT. Because food insecurity was the most significant problem for women with PD in the formative work, the investigators believe interventions will be most effective if couples can also engage in problem-solving around nutrition, meal preparation, and access to food.

The investigators propose to build on the World Health Organization (WHO) Problem Management Plus (PM+) intervention, which is based on problem-solving therapy (PST) and is effective at reducing depressive symptoms with individuals. PM+ has been adapted for the Malawi context and is currently undergoing an implementation evaluation. The investigators will adapt PM+ for couples with the goal of engaging partners to provide social support for PD, helping women brainstorm and solve problems around PD, food insecurity, and PMTCT adherence, and improving couple communication skills to help couples talk constructively about depression, nutrition and other needs, relationship challenges, and adherence to PMTCT.

ELIGIBILITY:
Inclusion Criteria:

* In a marriage or cohabitating union for at least 6 months.
* One member of the couple is a woman in the second or third trimester of pregnancy who is living with HIV and screens positive for depression (>10 on the PHQ9).
* Have revealed their HIV status to their partner if living with HIV>

Exclusion Criteria:

* Fear their safety would be at risk.
* Report incidents of severe intimate partner violence (IPV) in the past three months using the WHO IPV measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Participation in the intervention | following the intervention period, an average of 5 months
  Proportion of couples who attend 75% and 100% of sessions.
Retention | through study completion, an average of 11 months
  Proportion of couples who complete the study follow-up surveys at 3 months post-partum and 6 months post-partum
Intervention fidelity | following the intervention period, an average of 5 months
  Study managers will listen to audio recordings of the intervention sessions and complete checklists to assess whether or not each session component was completed.
Acceptability | Assessed at the 3-month post-partum follow-up
  Proportion of couples who report satisfaction with the intervention and proportion who would recommend the intervention to friends and neighbors

SECONDARY OUTCOMES:
Perinatal depression | 3 months post partum
  Using the Center for Epidemiologic Studies Depression Scale (CES-D scale), which is validated for people living with HIV in SSA. Scores range from 0 to 60 with higher scores indicating more depression symptomatology.
Perinatal depression | 6 months post-partum
  Using the Center for Epidemiologic Studies Depression Scale (CES-D scale), which is validated for people living with HIV in SSA. Scores range from 0 to 60 with higher scores indicating more depression symptomatology.
Perinatal viral suppression | 6 months post-partum
  This is a component of PMTCT. The lab at Zomba Central Hospital will use plasma samples to measure viral load.
Perinatal adherence to ART | 3 months post-partum
  This is a component of PMTCT. Using the Visual Analog Scale (VAS), women will report the proportion of prescribed ART doses taken during pregnancy and postpartum. Adherence will be defined as taking 100% of the prescribed medication during each time period.
Perinatal adherence to ART | 6 months post-partum
  This is a component of PMTCT. Using the Visual Analog Scale (VAS), women will report the proportion of prescribed ART doses taken during pregnancy and postpartum. Adherence will be defined as taking 100% of the prescribed medication during each time period.
Adherence to infant prophylaxis | 3 months post-partum
  This is a component of PMTCT. Women will be asked if they ingested Nevirapine (NVP) during labor and delivery (yes or no). Using the Visual Analog Scale (VAS), women will estimate adherence to NVP prophylaxis for the infant postpartum. Higher scores indicated better adherence.
Infant HIV testing | 3 months post-partum
  This is a component of PMTCT. Women will self-report whether they tested their infant for HIV after 8 weeks and the result of test (to be confirmed with medical records).
Breast feeding | 3 months post-partum
  This is a component of adherence to PMTCT. Women will be asked, "Are you currently exclusively breastfeeding your baby?"
Breast feeding | 6 months post-partum.
  This is a component of adherence to PMTCT. Women will be asked, "Are you currently exclusively breastfeeding your baby?"

CONTACTS AND LOCATIONS:
Overall Officials: Amy Conroy, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Invest in Knowledge (IKI), Zomba, Malawi

IPD SHARING:
Plan to Share IPD: Yes
The dataset will include self-reported demographic and behavioral data from surveys and laboratory data from blood specimens. Individual-participant level or IPD data will be shared. The data will be made in a de-identified format. In addition to the IPD dataset, the researcher will share the data dictionary and final protocol with amendments.
  Identifiable data will be de-identified prior to repository submission. All participant-level data will be preserved and shared through deposition in the NIMH Data Archive (NDA), a controlled access public repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All collection data will be shared automatically two years after the grant end date specified on the first Notice of Award. Any subject-level data and the associated analyzed data used in a journal publication will be shared at the time of publication, even if the publication occurs before the two-year automatic share date.
Access Criteria: The data will be made available for sharing with the general research community via the NDA website. Investigators at institutions with a Federal Wide Assurance (FWA) will be able to gain access to NDA data by submitting a data access request in accordance with applicable NDA policies. Data requests will be reviewed and granted by an NDA Data Access Committee. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.

REFERENCES:
- [Background] Bengtson AM, Filipowicz TR, Mphonda S, Udedi M, Kulisewa K, Meltzer-Brody S, Gaynes BN, Go VF, Chibanda D, Verhey R, Hosseinipour MC, Pence BW. An Intervention to Improve Mental Health and HIV Care Engagement Among Perinatal Women in Malawi: A Pilot Randomized Controlled Trial. AIDS Behav. 2023 Nov;27(11):3559-3570. doi: 10.1007/s10461-023-04070-8. Epub 2023 Apr 21. PMID 37084104
- [Background] Ramchandani P, Stein A, Evans J, O'Connor TG; ALSPAC study team. Paternal depression in the postnatal period and child development: a prospective population study. Lancet. 2005 Jun 25-Jul 1;365(9478):2201-5. doi: 10.1016/S0140-6736(05)66778-5. PMID 15978928
- [Background] Tuthill EL, Neilands TB, Johnson MO, Sauceda J, Mkandawire J, Conroy AA. A Dyadic Investigation of Relationship Dynamics and Depressive Symptoms in HIV-Affected Couples in Malawi. AIDS Behav. 2019 Dec;23(12):3435-3443. doi: 10.1007/s10461-019-02583-9. PMID 31273489
- [Background] Coleman SF, Mukasakindi H, Rose AL, Galea JT, Nyirandagijimana B, Hakizimana J, Bienvenue R, Kundu P, Uwimana E, Uwamwezi A, Contreras C, Rodriguez-Cuevas FG, Maza J, Ruderman T, Connolly E, Chalamanda M, Kayira W, Kazoole K, Kelly KK, Wilson JH, Houde AA, Magill EB, Raviola GJ, Smith SL. Adapting Problem Management Plus for Implementation: Lessons Learned from Public Sector Settings Across Rwanda, Peru, Mexico and Malawi. Intervention (Amstelveen). 2021 Jan-Jun;19(1):58-66. Epub 2021 Mar 31. PMID 34642580